CLINICAL TRIAL: NCT01221714
Title: Toxicity and Safety Evaluation of an Omega-3 Fatty Acid and a Multivitamin and Antioxidant Nutritional Preparation
Status: Terminated | Type: Observational
Why Stopped: Ameriscience went bankrupt.
Sponsor: AmeriSciences LP (Industry)
Collaborators: Bio-Medical Consultants, Inc. (Industry); Vantage Data Solutions Inc. (Industry); Esoterix, Inc. (Industry); Dr. Marwan Sabbagh, Study Monitor (Unknown)
Responsible Party: Carlos A. Montesinos/Director of Quality and Product Development, AmeriSciences
Other Study IDs: AS08-001
Record Dates: First submitted 2010-10-14; First posted 2010-10-15 (Estimated); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Healthy
Keywords: nutritional supplements; supplements; vitamins; omega-3; Amerisciences; Carlos Montesinos

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be drawn at baseline and three months to monitor hematology, blood chemistry, and urinalysis values for major changes. CBC, Chem-17, uric acid, lipid panel, PT/PTT, and urinalysis will be evaluated under fasting conditions.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Active/Placebo: ACTIVE VITAMIN; PLACEBO OMEGA MAX
- Active/Active: ACTIVE VITAMIN; ACTIVE OMEGA MAX
- Placebo/Active: PLACEBO VITAMIN; ACTIVE OMEGA MAX
- Placebo/Placebo: PLACEBO VITAMIN; PLACEBO OMEGA MAX

SUMMARY:
To evaluate the safety and tolerability of two supplements in healthy subjects taken daily for six months.

DETAILED DESCRIPTION:
The Lyndon B. Johnson Space Center (JSC) of the National Aeronautics and Space Administration (NASA) and AmeriSciences have entered into a Space Act Agreement (1), the primary objectives of which are the development of nutritional products in the form of dietary supplements to maintain homeostasis, and as countermeasures to reduce the biological effects and damages of long-duration spaceflight mediated through oxidative stress both in low Earth Orbit and planetary exploration of the solar system, as well as to provide optimal nutritional supplementation to aid in pre-spaceflight conditioning.

NASA has determined through pre-, in-, and post-flight assessment of cells, animals and humans that spaceflight induces oxidative stress on crewmembers. There are multiple potential sources of oxidative injury to include, but not limited to space radiation, noise, fuel reaction products, planetary regolith, and exercise. Furthermore, NASA has also determined that several foreseen and unforeseen physiological events can be controlled, avoided, or encouraged by means of dietary modification through supplements. Due to unforeseen limitation in the available fresh food supply for envisioned exploratory missions, it is desirable for NASA to have nutritional supplementation available to provide crewmembers with augmentation for the intrinsic defense systems against oxidative damage, as well as for potential nutritional contingencies such as food shortages and optimization of the diet. NASA has identified the need for specific micronutrient formulations to complement natural food sources, for astronaut protection during long-duration space flight.

AmeriSciences is a nutritional company that specializes in science-based product formulation, manufacturing under Good Manufacturing Practices (GMP) using standards modeled after those used by the pharmaceutical industry. It has been charged with the co-development, aid, clinical evaluation, construction, and production of said micronutrient formulations, to the level of specifications required to meet NASA's expectations for safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

To be eligible, patients must meet the following eligibility criteria:

1. Male or Female subject between the ages of 21 and 65 years
2. Capable of providing informed consent
3. Patients currently taking HMG-CoA reductase inhibitors (i.e. "statin" drugs), or any other drug known to interfere with serum transaminase (i.e. liver enzymes), must have history of stable liver function test since first taking such drugs.
4. Patients who usually and customarily take dietary supplements, including vitamins, must undergo a two-week washout period

Exclusion Criteria:

To be eligible, patients must not meet any of the following exclusion criteria:

1. Exposure to any investigational drug within 90 days of the beginning of this study
2. Known human immunodeficiency virus (HIV) seropositivity or Acquired Immunodeficiency Syndrome (AIDS); history of Hepatitis B (HBV), Hepatitis C (HCV) vital infection, unexplained elevated serum transaminase, or other hepatic disease. NOTE: HIV, HCV and HBV testing will not be performed as part of screening.
3. History of cancer within the last 5 years, except for basal or squamous cell cancer.
4. Allergy to fish (specifically sardines, anchovies or mackerel) or any of the investigational product components
5. Concomitant use, or use within less than a two-week period, of any other dietary supplement
6. Concomitant use of any drug known to interfere with laboratory measures such as:

   1. Niaspan (extended release niacin)
   2. Lamisil (terbinafine HCl)
   3. Chronic use of acetaminophen (>1,500 mg/day) (occasional use for minor aches and pains is excluded from this restriction)
   4. New prescriptions (< 90days) of HMG-CoA reductase inhibitors ("statins"), or patients currently on statins who have previously shown evidence of elevated serum transaminases
7. Currently diagnosed with multiple sclerosis, systemic lupus erythematosis, or other autoimmune disorders known to interfere with laboratory measures
8. Pregnancy, Lactation, or females actively attempting to become pregnant
9. History of alcoholism or drug abuse, unless it is determined that such past use would not influence laboratory measures (DSN4 criteria)
10. Any other active disease of a life-threatening nature or laboratory abnormality that, in the judgment of the investigator, may interfere with the interpretation, or increase risk of patient participation
11. Conditions that require nutritional therapy, such as:

    1. Pernicious anemia
    2. Iron-deficiency anemia
    3. Hartnup Disease or Pellagra
    4. Scurvy
    5. Beriberi-induced Endemic Neuritis

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Approximately 160-200 healthy volunteers at five to six study centers (25-50) per center) will be evaluated.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2010-10; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Montesinos, Principal Investigator — AmeriSciences LP
Locations (3):
- United States (3):
  - Mississippi Family Doctors, Pearl, Mississippi
  - Carolina Medical Associates, Charlotte, North Carolina
  - Logan General Hospital, Logan, West Virginia